CLINICAL TRIAL: NCT03418779
Title: Treatment Effects of Chinese Medicine (Yi-Qi-Qing-Jie Herbal Compound) Combined With Immunosuppression Therapies in IgA Nephropathy Patients With High-risk of End-stage Renal Disease (TCM-WINE)
Brief Title: Treatment Effects of Chinese Medicine (Yi-Qi-Qing-Jie Herbal Compound) Combined With Immunosuppression Therapies in IgA Nephropathy Patients With High-risk of ESRD
Acronym: TCMWINE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Shen, Professor & MD., Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCMWINE
Record Dates: First submitted 2018-01-11; First posted 2018-02-01 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: IgA Nephropathy at High Risk of Developing ESRD
Keywords: IgA nephropathy; immunosuppressive therapy; Yi-Qi-Qing-Jie herbal compound; high-risk IgAN; traditional chinese medicine
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Immunosuppressive Agents; Prednisolone; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and all other members with clinical involvement in the trial will be blinded to the treatment assignment for the duration of the trial. Relevant personnel have clear divisions of labor and strict permission restrictions. The blinding will be removed only if a participant has severe side effects that the affected participant will be withdrawn.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Experimental): Optimized supportive care, YQF placebo (oral granule), immunosuppression therapy comprises oral prednisolone plus intravenous cyclophosphamide.
  Interventions: Drug: Immunosuppressants; Other: Optimized Supportive Care; Other: Yi-Qi-Qing-Jie herbal compound placebo
- YQF Group (Experimental): Optimized supportive care, YQF (oral granule), immunosuppression therapy comprises oral prednisolone plus intravenous cyclophosphamide.
  Interventions: Drug: The Yi-Qi-Qing-Jie herbal compound; Drug: Immunosuppressants; Other: Optimized Supportive Care

INTERVENTIONS:
Drug: The Yi-Qi-Qing-Jie herbal compound — The compounds are blends of individual herbal extracts from YQF (consisting of Astragalus membranaceus, Saposhnikovia divaricata (turcz.) Schischk, Flos lonicerae, Angelica sinensis, Dioscorea nipponica, Hedyotis diffusa Willd, rhubarb, Spatholobus suberectus, with the effect of reinforcing Qi and activating blood, clearing away heat and poison, dissolving dampness and downbearing turbid) dissolved in 150 ml boiled water and taken orally twice a day for the duration of the treatment and follow-up phases.
  Arms: YQF Group
Drug: Immunosuppressants — Immunosuppression therapy comprises oral prednisolone (0.5-0.8 mg/kg/day; exact dose decided by the investigator, maximum dose not exceeding 60 mg/day) for 8 weeks, then tapered by 5-10 mg/day every 4 weeks, with a total treatment period of 24-32 weeks. Participants with persistent proteinuria ≥ 1 g/day after 8 weeks of corticosteroid monotherapy will receive 0.8-1.0 g of intravenous cyclophosphamide (CTX) every 4 weeks, total dose of not exceeding 8 g (exact dose decided by the site investigator). If severe CTX-related adverse events occur, such as alanine transaminase (ALT) exceeding the upper limit of two times, infections requiring hospitalization, granulocytes < 3.0 × 109/L and platelets < 50.0 × 109/L, CTX will stop being administered, symptoms will be treated, and adverse events recorded. Also, the frequency of detection will be increased to once every 2 weeks and the affected participant will be withdrawn if persistent infection or myelosuppression occurs.
  Other Names: prednisolone; cyclophosphamide
Other: Optimized Supportive Care — The optimized supportive care included:
  1. Lifestyle: low-salt, restricted protein dietary with sufficient calorie supply, smoking cessation, moderate alcohol consumption and keeping a healthy weight
  2. The use of renin-angiotensin system blockade: lowering blood pressure to a target below 135/85 mmHg, during which treatment was adjusted to ensure that patients were receiving the maximum labelled or tolerated dose of RAS blockade
  3. Patients with Diabetes Mellitus received insulin or oral hypoglycemic agents to achieve HbA1c≤ 7.0%
  4. Received uricosuric agents or xanthine oxidase inhibitors as necessary to achieve serum uric acid <6 mg/dL in female, <7 mg/dL in male
Other: Yi-Qi-Qing-Jie herbal compound placebo — Patients will receive Yi-Qi-Qing-Jie herbal compound placebo instead for the duration of the treatment and follow-up phases. The major component of the placebo is malt dextrin which looks, smells and tastes like YQF compound, and it comes in packaging with a similar appearance to YQF compound; it is also dissolved in 150 ml boiled water and taken orally twice a day.
  Arms: Control Group

SUMMARY:
The TCM-WINE study is a single-center, prospective, double-blind randomized placebo-controlled trial. Based on optimal supportive care, the trial is aiming to assess superiority with regard to renal protection and reduction of severe treatment-related adverse events of Yi-Qi-Qing-Jie formula (YQF) combined therapy compared with immunosuppression monotherapy in high-risk IgAN.

DETAILED DESCRIPTION:
The investigators plan to randomize 60 participants with biopsy-proven IgAN to a YQF combined group (YQF compound combined with prednisolone, and cyclophosphamide if necessary) or an immunosuppression group (placebo-YQF combined with prednisolone, and cyclophosphamide if necessary). The two groups will enter a 48-week in-trial treatment phase and receive post-trial follow-up until 50% (30/60) have a composite endpoint or have been followed for 3 years (study completion). All patients will receive optimal supportive care.

ELIGIBILITY:
Inclusion Criteria:

1. patients who maintain regular follow-ups at Guang'anmen Hospital, agree to participate, and provide informed consent;
2. biopsy-proven IgA nephropathy, with recent progression to high-risk IgAN*;
3. eGFR 15 to 60 ml/min/1.73 m2, calculated with the use of CKD-EPI Creatinine Equation 2009.

   * High-risk IgAN: persistent proteinuria ≥ 1 g/d despite at least 8 weeks of optimal supportive care [maximally tolerated RAS blocker which refers to no symptomatic hypotension, no hyperkalemia, and serum creatinine increased by not more than 30% of baseline, blood pressure control meeting targets (135/85 mmHg or lower), and dietary management (sodium intake less than 6 g/d, protein intake of 0.6-0.8 g/kg/day, and low-fat diet)], the mean annual eGFR decline rate (eGFR-slope) >10 ml/min per 1.73 m2 per year, while needing to restart immunosuppressive therapy; or eGFR<60 ml/min/1.73 m2 at the first diagnosis.

Exclusion Criteria:

1. secondary IgAN;
2. comorbidity of other primary or secondary glomerular diseases;
3. comorbidity of severe primary diseases such as cardiovascular, hepatic, cerebral, and hematopoietic system diseases or mental disorders;
4. allergy or intolerance to the experimental medication (e.g., RAS blockers, prednisolone, cyclophosphamide, YQF compound and its placebo compound);
5. contraindications to immunosuppression therapy-acute and chronic infectious diseases, malignancies, leukopenia, thrombocytopenia, gastrointestinal hemorrhage, ulcers of stomach or duodenum, post-transplantation;
6. pregnant or lactating women;
7. unwilling to participate in this study, failure to accept or tolerate Chinese medicine compound;
8. history of alcohol or drug abuse;
9. poor compliance, loss to follow-up;
10. participation in another clinical investigation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
First occurrence of 40% decrease in eGFR from baseline | Baseline, until the first occurrence or 3 years
First occurrence of progression to continuous renal replacement | Until occurrence or 3 years
Death due to renal disease | Until occurrence or 3 years

SECONDARY OUTCOMES:
Mean annual reduction in eGFR based on SCr | 48 weeks
  eGFR slope
Proteinuria remission | Week 24, 36, and 48 in the treatment period, and month 6, 12, 24, or 36 if possible
  Prescribed as proteinuria < 0.5 g/day
The remission rate of symptoms and inflammation status | Week 48
  The subjective symptoms and inflammation status will be scored on a four-point scale ranging from 0 (absent) to 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Study Chair — Guang anmen Hospital, China Academy of Chinese Medical Sciences
Locations (1):
- Guang anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Li S, Li JP. Treatment effects of Chinese medicine (Yi-Qi-Qing-Jie herbal compound) combined with immunosuppression therapies in IgA nephropathy patients with high-risk of end-stage renal disease (TCM-WINE): study protocol for a randomized controlled trial. Trials. 2020 Jan 6;21(1):31. doi: 10.1186/s13063-019-3989-9. PMID 31907076